CLINICAL TRIAL: NCT05445557
Title: A Double-Blind, Placebo-Controlled Phase Followed by An Open-Label Phase to Evaluate the Safety and Efficacy of RZL-012 in Subjects Seeking Fat Reduction in the Flanks
Brief Title: Evaluation of Safety and Efficacy of RZL-012 in Subjects Seeking Fat Reduction in the Flanks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Raziel Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RZL-012-FL-P2US-001
Record Dates: First submitted 2022-02-14; First posted 2022-07-06 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-02

CONDITIONS: Flank Mass
MeSH Terms: interventions — RZL-012

STUDY DESIGN:
Intervention Model Description: Each of the subject's flanks will be randomized for RZL-012 and placebo injections.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RZL-012 50mg/ml (Active Comparator): Subjects flanks treated with RZL-012 (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal doses 412.5 mg. Each injection point will be dosed with 7.5 mg for in a volume of 0.15 mL/injection site.
  Interventions: Drug: RZL-012
- Placebo (Placebo Comparator): Subjects flanks treated with placebo (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal volume of 8.25mL. Each injection point will be dosed with 0.15 mL/injection site.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RZL-012 — small synthetic molecule for submental fat reduction
  Arms: RZL-012 50mg/ml
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A total of 12 subjects will be injected with RZL-012 and placebo. Each of the subject's flanks will be randomized for each of the treatment. A total of 24 flanks will be randomized in the double blind phase. They will be monitored for safety and efficacy for 12 weeks. After codes opening, a second treatment cycle on the previously untreated contralateral flank will be done. Subjects will be monitored for safety and efficacy for additional 12 weeks.

DETAILED DESCRIPTION:
This clinical trial is comprised of a double-blind, placebo-controlled phase followed by an open-label phase.

The double-blind, placebo-controlled phase of the trial will consist of a screening period, baseline visit and a 12-week post-treatment follow-up period. At the baseline visit, each flank (right and left) of each study participant will be randomized into either the active RZL-012 treatment group or the placebo group and each flank will receive multiple injections in a single session of RZL-012 or placebo. Blood samples will be collected for 6 of the 12 subjects for PK analyses. All subjects will be followed up for 12 weeks after the single treatment session.

Upon completion of the double-blind phase of the study, and the opening of codes subjects will be offered RZL-012 open-label treatment in the flank previously treated with placebo. Consenting subjects will be followed for safety and efficacy for an additional 12 weeks.

In both the double-blind and open-label phases of the study, subjects will be monitored for adverse events (AEs). Subjects will return to the site for visits at 1 week, 4 weeks, 8 weeks, and 12 weeks post treatment and will be monitored for safety and efficacy during these visits.

Subjects who will be collected with PK will return to the clinic at Day 1 post injection for further PK samples.

The dimensions of flanks will be measured using 3D images and volumetric calculations using Canfield 3D images.

ELIGIBILITY:
Inclusion Criteria:

* Is a male or female subject between the ages of 18 and 65 years, inclusive.
* Has body mass index (BMI) BMI of ≥ 22 and < 30.
* Has clearly visible and palpable fat in the flanks
* Has symmetrical appearance of right and left flanks
* Agrees to maintain weight (i.e., within 5% of body weight) by not making any changes in diet.
* Agree to avoid exposure of the treated area to the sun for at least 1 month after each treatment session.
* If female, is not pregnant or breastfeeding based on the following:

  1. agree to the use of highly effective contraceptive methods for at least 2 weeks before baseline until 28 days after the last day of study drug and a negative urine pregnancy test at screening and baseline; or
  2. is of nonchildbearing potential defined as clinically infertile as the result of surgical sterilization (hysterectomy, bilateral tubal ligation, and/or bilateral oophorectomy); or
  3. is confirmed postmenopausal status (defined as either having amenorrhea for ≥ 12 consecutive months without another cause, having documented serum follicle-stimulating hormone (FSH) level > 40 mIU/mL, or having another documented medical condition (e.g., was born without a uterus))
* If male (with or without vasectomy), agree to the use of highly effective contraceptive methods, e.g. condom, from study baseline until 7 days after the last day of study drug.
* Is willing to avoid strenuous exercise for seven (7) days post treatment.
* Is motivated to adhere to the visit schedule and protocol requirements.
* Is willing and able to sign an Institutional Review Board (IRB) approved informed consent form (ICF) indicating that they are aware of the investigational nature of the study.

Exclusion Criteria:

* Is unable to tolerate subcutaneous injections.
* Has dysfunctional gallbladder activity (e.g., underwent cholecystectomy or cholecystitis).
* Has an uncontrolled systemic disease that is not stabilized (i.e., cardiovascular disease, mental illness).
* Has used anticoagulation therapies that may increase bleeding or bruising (i.e., aspirin, ibuprofen, vitamins, and herbal preparations) for seven (7) days prior to treatment.
* Has medication or a history of coagulopathy.
* Has a history or family history of venous thrombotic disease.
* Had a non-invasive fat reduction and/or body contouring procedure in the flanks within the past 12 months.
* Has any scars, unshaven hair, tattoos, on or near the proposed treatment area.
* Has significant history or current evidence of a medical, psychological or other disorder that, in the Investigator's opinion, would preclude enrollment in the study.
* Has an active dermatitis or open wound in the proposed treatment area.
* Abnormal coagulation profile including: activated partial thromboplastin time (aPTT) > ULN, international normalized ratio (INR) > ULN reference range (> 1.3), prothrombin time (PT) > ULN.
* Has an active bacterial, fungal, or viral infection in the proposed treatment area.
* Has known allergic reactions to any injectables.
* Has been treated chronically in the past 3 months prior to study entry with systemic steroids or immunosuppressive drugs.
* Has been treated chronically at least one (1) week prior to study entry with non-steroidal anti-inflammatory drugs (NSAIDs).
* Current participation or participation within three (3) months prior to the start of this study in a drug or other investigational research study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luxurgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: flanks
Groups:
- All Study Participants: Subjects flanks treated with RZL-012 (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal doses 412.5 mg. Each injection point will be dosed with 7.5 mg for in a volume of 0.15 mL/injection site.
  RZL-012: small synthetic molecule for submental fat reduction
Period: Double Blind Part
Arm/Group | All Study Participants
Started (RZL-012) | 12; 24 flanks
Flanks Treated With RZL-012 | 12; 12 flanks
Flanks Treated With Placebo | 12; 12 flanks
Completed | 11; 22 flanks
Not Completed | 1; 2 flanks
Not completed — Lost to Follow-up | 1
Period: Open Label - Active Only
Arm/Group | All Study Participants
Started | 9; 9 flanks
Completed | 9; 9 flanks
Not Completed | 0; 0 flanks

BASELINE CHARACTERISTICS:
Groups:
- RZL-012 50mg/ml or Placebo: Subjects flanks treated with RZL-012 (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal doses 412.5 mg. Each injection point will be dosed with 7.5 mg for in a volume of 0.15 mL/injection site.
  RZL-012: small synthetic molecule for submental fat reduction
  Subjects flanks treated with placebo (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal volume of 8.25mL. Each injection point will be dosed with 0.15 mL/injection site.
  Placebo: Placebo
Arm/Group | RZL-012 50mg/ml or Placebo
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The results from the double blind phase and open label phase are presented. The number of subjects that continued to the open label phase were 9.
  years
    Double blind phase | 43 (12.2)
    Open Label phase: number analyzed (Participants) | 9
    Open Label phase | 44.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The results from the double blind phase are presented together with the results from the open label phase.
  Only 9 subjects continued to the open label phase
  Participants
    Double blind phase: Female | 10
    Double blind phase: Male | 2
    Open Label phase: number analyzed (Participants) | 9
    Open Label phase: Female | 7
    Open Label phase: Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: he results from the double blind phase are presented together with the results from the open label phase.
  Only 9 subjects continued to the open label phase
  Participants
    Double Blind phase: American Indian or Alaska Native | 0
    Double Blind phase: Asian | 0
    Double Blind phase: Native Hawaiian or Other Pacific Islander | 0
    Double Blind phase: Black or African American | 2
    Double Blind phase: White | 10
    Double Blind phase: More than one race | 0
    Double Blind phase: Unknown or Not Reported | 0
    Open label phase: number analyzed (Participants) | 9
    Open label phase: American Indian or Alaska Native | 0
    Open label phase: Asian | 0
    Open label phase: Native Hawaiian or Other Pacific Islander | 0
    Open label phase: Black or African American | 1
    Open label phase: White | 8
    Open label phase: More than one race | 0
    Open label phase: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events [AEs]
Description: Safety
Time Frame: 12 weeks for the Double-Blind Phase and 12 weeks for the Open-Label Phase
Population: The data for double blind and open label phase are presented. A total of 9 subjects continued to open label phase.
Measure: Number; unit: participants
Groups:
- Placebo: Subjects flanks treated with placebo (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal volume of 8.25mL. Each injection point will be dosed with 0.15 mL/injection site.
  Placebo: Placebo
  RZL-012: small synthetic molecule for submental fat reduction
- RZL-012 Open Label: Subjects that were treated with placebo in their flanks chose to treat these flanks with RZL-012
Arm/Group | RZL-012 50mg/ml | Placebo | RZL-012 Open Label
Number analyzed (Participants) | 12 | 12 | 9
participants
  AE Related Study Treatment | 12 | 12 | 9
  Related to Injection Procedure | 12 | 12 | 9
  Severe Adverse Events | 0 | 0 | 0

2. Secondary Outcome: Efficacy - Number of Flanks That Have Change in Score According Physician Global Assessment Scale
Description: To compare the proportion of flanks having an improvement as indicated by reduction in score from 6 to 0 according to the Physician Global Assessment Scale (GAIS) in RZL-01-treated flanks vs placebo-treated flanks
Time Frame: 12 weeks for the Double-Blind Phase and 12 weeks for the Open-Label Phase
Population: A total of 9 subjects continued to the open label phase
Measure: Number; unit: flanks
Units Other Than Participants: Flanks
Groups:
- RZL-012 50mg/ml Double Blind: Subjects flanks treated with RZL-012 (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal doses 412.5 mg. Each injection point will be dosed with 7.5 mg for in a volume of 0.15 mL/injection site.
  RZL-012: small synthetic molecule for submental fat reduction
- Placebo Double Blind: Subjects flanks treated with PLACEBO (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 . Each injection point will be dosed with of 0.15 mL/injection site.
  Placebo: Vehicle of drug product
- RZL-012 Open Label Treatment: Subjects flanks treated with RZL-012 (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal doses 412.5 mg. Each injection point will be dosed with 7.5 mg for in a volume of 0.15 mL/injection site.
Arm/Group | RZL-012 50mg/ml Double Blind | Placebo Double Blind | RZL-012 Open Label Treatment
Number analyzed (Participants) | 11 | 11 | 9
Number analyzed (Flanks) | 11 | 11 | 9
flanks
  Marked Improvement | 7 | 0 | 0
  Moderate Improvement | 2 | 0 | 0
  Slight Improvement | 1 | 0 | 7
  No Change | 1 | 11 | 2

3. Secondary Outcome: Efficacy - Change in Satisfaction Score
Description: To compare the proportion of subjects who are satisfied with treatment results as indicated by a binary yes/no satisfaction questionnaire in RZL-012-treated flanks vs placebo-treated flanks
Time Frame: 12 weeks for the Double-Blind Phase and 12 weeks for the Open-Label Phase
Population: A total of 9subjects continued to the open label phase
Measure: Count of Participants; unit: Participants
Groups:
- RZL-012 50mg/ml or Placebo: Subjects flanks treated with RZL-012 (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal doses 412.5 mg. Each injection point will be dosed with 7.5 mg for in a volume of 0.15 mL/injection site.
  Subjects flanks treated with placebo (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal volume of 8.25mL. Each injection point will be dosed with 0.15 mL/injection site.
  Placebo: Placebo
  RZL-012: small synthetic molecule for submental fat reduction
Arm/Group | RZL-012 50mg/ml or Placebo
Number analyzed (Participants) | 11
Participants
  RZL-012 - Double blind phase: Satisfied | 9
  RZL-012 - Double blind phase: Not Satisfied | 2
  Placebo Double blind phase: Satisfied | 1
  Placebo Double blind phase: Not Satisfied | 10
  RZL-012 Open Label phase: number analyzed (Participants) | 9
  RZL-012 Open Label phase: Satisfied | 6
  RZL-012 Open Label phase: Not Satisfied | 3

4. Secondary Outcome: Efficacy - Relative Change in Measured Fat Volume
Description: Measure the relative mean reduction in volume (%) at post treatment vs. baseline for each of the treated flanks, as measured by 3D images using the Canfield 3D system in RZL-012-treated flanks vs placebo-treated flanks at 12 weeks vs. baseline
Time Frame: 12 weeks for the Double-Blind Phase and 12 weeks for the Open-Label Phase. Baseline for the open-label phase considered to be 12 weeks after double blind treatment
Population: A total of 9 subjects continued to the open label phase
Measure: Mean (Standard Deviation); unit: percentage of change from baseline.
Units Other Than Participants: Flanks
Groups:
- RZL-012 50mg/ml Double Blind Part; RZL-012 Open Label Part: Subjects flanks treated with RZL-012 (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal doses 412.5 mg. Each injection point will be dosed with 7.5 mg for in a volume of 0.15 mL/injection site.
  RZL-012: small synthetic molecule for submental fat reduction
- Placebo Double Blind Part: Subjects flanks treated with placebo (in the double blind phase) will undergo a single treatment session with 50-55 injections. The maximal number of injections will be 55 with maximal volume of 8.25mL. Each injection point will be dosed with 0.15 mL/injection site.
  Placebo: Placebo
Arm/Group | RZL-012 50mg/ml Double Blind Part | Placebo Double Blind Part | RZL-012 Open Label Part
Number analyzed (Participants) | 11 | 11 | 9
Number analyzed (Flanks) | 11 | 11 | 9
percentage of change from baseline. | -37 (55.2) | 33 (41.4) | -48.9 (65.9)

5. Secondary Outcome: Efficacy -Number of Participant With Correct Identification by Reviewers
Description: Blinded reviewers will identify, per patient, the flank treated with test compound (active) vs the flank treated with Placebo. Success will be defined as at least 70% correct identification vs the expected 50% correct identification based on random guessing
Time Frame: 12 weeks 12 weeks for the Double-Blind Phase
Measure: Count of Participants; unit: Participants
Arm/Group | RZL-012 50mg/ml
Number analyzed (Participants) | 11
Participants
  Reviewer 1 - Correct identification of active treated flanks | 5
  Reviewer 2 - Correct identification of active treated flanks | 6

6. Secondary Outcome: Pharmacokinetics Measure - Drug Concentration in the Blood (ng/mL)
Description: Measurement of maximum drug concentration (Cmax) (ng/mL) in the blood
Time Frame: 30 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | RZL-012 50mg/ml
Number analyzed (Participants) | 6
ng/ml | 961.8 (273.4)

ADVERSE EVENTS:
Time Frame: 12 weeks Double blind phase and 12 weeks open label phase
Arm/Group | RZL-012 50mg/ml | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | RZL-012 50mg/ml (N=12) | Placebo (N=12)
edema (General disorders) | 11 | 12 — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
pain (General disorders) | 12 | 12 — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
tenderness (General disorders) | 4 | 1 — GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS
Hypoesthesia (Nervous system disorders) | 5 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 6 | 8
erythema (Skin and subcutaneous tissue disorders) | 7 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 7
edema Open Label phase (General disorders) | 9/9 | 0
pain open label phase (General disorders) | 9/9 | 0
Tenderness - Open Label phase (General disorders) | 2/9 | 0
Hypoesthesia Open Label phase (Nervous system disorders) | 7/9 | 0
Erythema open label phase (Skin and subcutaneous tissue disorders) | 7/9 | 0
Pruritus Open Label phase (Skin and subcutaneous tissue disorders) | 2/9 | 0
Skin Hyperpigmentation open label phase (Skin and subcutaneous tissue disorders) | 3/9 | 0
Skin irritation Open Label phase (Skin and subcutaneous tissue disorders) | 1/9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT05445557/Prot_001.pdf
  • Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT05445557/SAP_002.pdf